CLINICAL TRIAL: NCT00004294
Title: Phase I Study of Retrovirally Mediated Transfer of the Human Glucocerebrosidase Gene Into Peripheral Blood Stem Cells for Autologous Transplantation in Patients With Type I Gaucher Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pittsburgh (Other)
Purpose: Treatment
Other Study IDs: 199/11727; UPITTS-GAUCHER
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Gaucher's Disease
Keywords: Gaucher's disease; inborn errors of metabolism; rare disease; sphingolipidoses
MeSH Terms: conditions — Gaucher Disease; Metabolism, Inborn Errors; Rare Diseases; Sphingolipidoses

INTERVENTIONS:
Genetic: human glucocerebrosidase gene into autologous peripheral blood stem cells

SUMMARY:
OBJECTIVES: I. Transfer the human glucocerebrosidase (GC) gene into peripheral blood stem cells (PBSC) obtained from patients with type I Gaucher disease using a retroviral vector.

II. Transplant the autologous transduced PBSC in these patients. III. Measure the carriage and expression of the transferred gene and its duration in peripheral blood leukocytes.

IV. Assess the clinical effects of transplanting genetically corrected PBSC.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo autologous transplantation using peripheral blood stems cells (PBSC) stimulated with filgrastim (G-CSF) and transduced with a retroviral vector containing the human glucocerebrosidase gene (R-GC). Patients may receive up to 4 transplants if a deficient glucocerebrosidase level is found in peripheral leukocytes 1 month following transplantation.

The G-CSF-stimulated PBSC are enriched for CD34-positive stem cells and transduced with the R-GC vector. Stem cells with normal gene activity are selected for transplantation.

Patients are followed every month for 6 months, every 6 months for 18 months, and then annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Enzyme proven type I Gaucher disease Glucocerebrosidase (GC) activity less than 30% of normal GC mutation identified Significant signs and symptoms of disease prior to therapy initiation At least 1 of the following after 12 months of therapy: Liver at least 2 times normal size Spleen at least 5 times normal size Platelet count greater than 150,000/mm3 Clinical bone disease with pain, fractures, or infarctions Multiple sites of marrow involvement Angiotensin-converting enzyme at least 1.5 times normal No GC antibody At least 3 of the following responses to therapy: Hemoglobin increase of 2 g/dL Platelet count increase of 50% Spleen or liver size decrease at least 25% Improvement in MRI or x-ray of the bones Nontartrate inhibitable acid phosphatase decrease of 50% Angiotensin-converting enzyme decrease of 50% OR Previously untreated and immediate enzyme therapy would not be life saving Meets at least 2 of the following criteria: Spleen at least 5 times normal size or liver at least 2 times normal size by physical exam and MRI Hemoglobin less than 11 g/dL Platelet count less than 90,000/mm3 Disabling bone pain with degenerative changes on x-ray Multiple sites of bone marrow infiltration and evidence of bony changes Pulmonary compromise with clubbing and PaO2 less than 70 mm Hg Biopsy proven cirrhosis and elevated hepatic parenchymal enzymes Bleeding esophageal varices --Prior/Concurrent Therapy-- At least 3 months since any prior investigational therapy Concurrent enzyme replacement therapy may be tapered on study --Patient Characteristics-- HIV negative No malignant disease No known sensitivity to egg or murine products Not pregnant or nursing Fertile patients must use effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: John Barranger, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States